CLINICAL TRIAL: NCT02957370
Title: Electro-Phage and Colorimetric Aptamer Sensors for Clinical Staging and Monitoring of Bladder Cancer
Brief Title: Molecular Biosensors for Detection of Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: HS#2014-1758
Record Dates: First submitted 2015-06-10; First posted 2016-11-07 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diagnosed Urinary Bladder Neoplasms: Patients who are being monitored for bladder cancer will be the experimental group to test the electro-phage and aptamer approach to following bladder cancer biomarkers
- Non-Urinary Bladder Neoplasms: Patients being treated for hematuria will provide a negative control to provide data from testing for biomarkers in patients being treated for other diseases.

SUMMARY:
This project focuses on developing specific and sensitive detectors of biomarker-based signatures associated with diagnosed and recurrent bladder cancer.

DETAILED DESCRIPTION:
The focus of this research is to discover urinary biomarker(s) that is distinct to bladder cancer, while developing molecular sensors that can detect the urinary anomalies. By applying in vitro selection techniques, both entities (biomarker discovery and sensor development) will be done simultaneously.

All patients with bladder cancer diagnosis undergoing transurethral resection bladder tumor (TURBT), those under surveillance for bladder cancer and patients presenting with microscopic and visible (gross) hematuria will be invited to participate in the study. Patients will undergo a standard of care evaluation as previously described (upper urinary tract imaging, cystouretheroscopy and urine testing with urinalysis, culture and cytology).

Urine samples (10 mL) for the study will be collected prior to initial cystoscopy and/or TURBT. The specimen will be barcoded and tracked by the UC Irvine Health software. Barcode encoding will ensure that the identity of the patient and his/her clinical outcome will not be available to the researchers for a blinded trial.

Patients involved in this study will only provide his or her urine for fundamental science research; beyond that, standard of care will be provided for the patients. With respect to the collected urine, it will be used as a medium for phage and aptamer production in an in vitro fashion. The generated molecular probes will be use to assess and elucidate biomarkers present for individuals with bladder cancer.

100 patients who are being monitored for bladder cancer will be the experimental group to test the electro-phage and aptamer approach to following bladder cancer biomarkers. Additionally, 100 patients being treated for hematuria will provide a negative control to provide data from testing for biomarkers in patients being treated for other diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Patients with diagnosed bladder cancer, undergoing transurethral resection bladder tumor (TRUBT), or under surveillance (within 2 years) for recurrent bladder cancer
* Patients with microscopic and macroscopic hematuria
* Willing and able to consent

Exclusion Criteria:

* Patients <18 years old
* Patients who are not able to give consent for study
* Patients with urinary diversions
* Patients who have had a recent percutaneous or endoscopic procedures for upper tract diseases such as stones or other conditions
* Patients who have ureteral stents placed for upper urinary tract obstruction
* Patients with recent trauma in kidney, bladder or perineal area, which may be the cause of hematuria
* Minors will be excluded from this study because ureteral stent placement is usually performed in adult patients. Additionally, minors are treated at CHOC Hospital, and not UCIMC.
* Women who are pregnant are excluded from this study since surgical treatments are not typically performed on pregnant women. Watchful waiting is the preferred approach for pregnant women. Furthermore, this research does not directly benefit the pregnant woman or fetus, and biomedical knowledge can be obtained using subjects who are not pregnant. Therefore, per the federal regulations, pregnant women will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited at the University of California, Irvine Medical Center Douglas Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2015-06-11 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Urinary "Fingerprint" for Urinary Bladder Neoplasms | Four Years
  A representative sequence from each class of the selected population will be synthesized and the fundamental properties for each aptamer sequences such as dissociation constant, switching performance, sensitivity, selectivity, and detection range will be measured using a Förster resonance energy transfer (FRET) system.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Landman, MD, Principal Investigator — UC Irvine
Locations (1):
- University of California Irvine, Orange, California, United States

REFERENCES:
- [Background] Kay, B. K. (1996) Table 15. M13 Stability and Instability, In Phage Display of Peptides and Proteins: A Laboratory Manual (Kay, B. K., Winter, J., McCafferty, J., Ed.), p 337, Academic Press, San Diego.
- [Background] Mohan K, Donavan KC, Arter JA, Penner RM, Weiss GA. Sub-nanomolar detection of prostate-specific membrane antigen in synthetic urine by synergistic, dual-ligand phage. J Am Chem Soc. 2013 May 22;135(20):7761-7. doi: 10.1021/ja4028082. Epub 2013 May 13. PMID 23614709
- [Background] Arter JA, Diaz JE, Donavan KC, Yuan T, Penner RM, Weiss GA. Virus-polymer hybrid nanowires tailored to detect prostate-specific membrane antigen. Anal Chem. 2012 Mar 20;84(6):2776-83. doi: 10.1021/ac203143y. Epub 2012 Mar 7. PMID 22339784
- [Background] Arter JA, Taggart DK, McIntire TM, Penner RM, Weiss GA. Virus-PEDOT nanowires for biosensing. Nano Lett. 2010 Dec 8;10(12):4858-62. doi: 10.1021/nl1025826. Epub 2010 Nov 1. PMID 21038915
- [Background] Diaz JE, Yang LM, Lamboy JA, Penner RM, Weiss GA. Synthesis of a virus electrode for measurement of prostate specific membrane antigen. Methods Mol Biol. 2009;504:255-74. doi: 10.1007/978-1-60327-569-9_16. PMID 19159102
- [Background] Donavan KC, Arter JA, Weiss GA, Penner RM. Virus-poly(3,4-ethylenedioxythiophene) biocomposite films. Langmuir. 2012 Aug 28;28(34):12581-7. doi: 10.1021/la302473j. Epub 2012 Aug 16. PMID 22856875
- [Background] Weiss GA, Penner RM. The Promise of Phage Display: Customized Affinity and Specificity. Anal Chem. 2008 May 1;80(9):3082-3089. doi: 10.1021/ac086009h. No abstract available. PMID 28193009
- [Background] Yang LM, Diaz JE, McIntire TM, Weiss GA, Penner RM. Direct electrical transduction of antibody binding to a covalent virus layer using electrochemical impedance. Anal Chem. 2008 Aug 1;80(15):5695-705. doi: 10.1021/ac8008109. Epub 2008 Jul 1. PMID 18590279
- [Background] Yang LM, Tam PY, Murray BJ, McIntire TM, Overstreet CM, Weiss GA, Penner RM. Virus electrodes for universal biodetection. Anal Chem. 2006 May 15;78(10):3265-70. doi: 10.1021/ac052287u. PMID 16689525
- [Background] Hanahan D, Weinberg RA. The hallmarks of cancer. Cell. 2000 Jan 7;100(1):57-70. doi: 10.1016/s0092-8674(00)81683-9. No abstract available. PMID 10647931
- [Background] Wallace TJ, Torre T, Grob M, Yu J, Avital I, Brucher B, Stojadinovic A, Man YG. Current approaches, challenges and future directions for monitoring treatment response in prostate cancer. J Cancer. 2014 Jan 1;5(1):3-24. doi: 10.7150/jca.7709. PMID 24396494
- [Background] Romero Otero J, Garcia Gomez B, Campos Juanatey F, Touijer KA. Prostate cancer biomarkers: an update. Urol Oncol. 2014 Apr;32(3):252-60. doi: 10.1016/j.urolonc.2013.09.017. Epub 2014 Feb 1. PMID 24495450
- [Background] Guan W, Duan X, Reed MA. Highly specific and sensitive non-enzymatic determination of uric acid in serum and urine by extended gate field effect transistor sensors. Biosens Bioelectron. 2014 Jan 15;51:225-31. doi: 10.1016/j.bios.2013.07.061. Epub 2013 Aug 7. PMID 23968728
- [Background] Yang LM, Diaz JE, McIntire TM, Weiss GA, Penner RM. Covalent virus layer for mass-based biosensing. Anal Chem. 2008 Feb 15;80(4):933-43. doi: 10.1021/ac071470f. Epub 2008 Jan 17. PMID 18198846
- [Background] Brigati JR, Petrenko VA. Thermostability of landscape phage probes. Anal Bioanal Chem. 2005 Jul;382(6):1346-50. doi: 10.1007/s00216-005-3289-y. Epub 2005 Jun 18. PMID 15965686
- [Background] Nanduri V, Sorokulova IB, Samoylov AM, Simonian AL, Petrenko VA, Vodyanoy V. Phage as a molecular recognition element in biosensors immobilized by physical adsorption. Biosens Bioelectron. 2007 Jan 15;22(6):986-92. doi: 10.1016/j.bios.2006.03.025. Epub 2006 May 30. PMID 16730970
- [Background] Zavada J, Zavadova Z, Zat'ovicova M, Hyrsl L, Kawaciuk I. Soluble form of carbonic anhydrase IX (CA IX) in the serum and urine of renal carcinoma patients. Br J Cancer. 2003 Sep 15;89(6):1067-71. doi: 10.1038/sj.bjc.6601264. PMID 12966427
- [Background] Huang S, Rhee E, Patel H, Park E, Kaswick J. Urinary NMP22 and renal cell carcinoma. Urology. 2000 Feb;55(2):227-30. doi: 10.1016/s0090-4295(99)00401-x. PMID 10688084
- [Background] Kaya K, Ayan S, Gokce G, Kilicarslan H, Yildiz E, Gultekin EY. Urinary nuclear matrix protein 22 for diagnosis of renal cell carcinoma. Scand J Urol Nephrol. 2005;39(1):25-9. doi: 10.1080/00365590410002500. PMID 15764267
- [Background] Myers-Irvin JM, Landsittel D, Getzenberg RH. Use of the novel marker BLCA-1 for the detection of bladder cancer. J Urol. 2005 Jul;174(1):64-8. doi: 10.1097/01.ju.0000162022.36772.a4. PMID 15947579
- [Background] van Rhijn BW, van der Poel HG, van der Kwast TH. Urine markers for bladder cancer surveillance: a systematic review. Eur Urol. 2005 Jun;47(6):736-48. doi: 10.1016/j.eururo.2005.03.014. Epub 2005 Mar 23. PMID 15925067
- [Background] Majumdar S, Hajduczki A, Mendez AS, Weiss GA. Phage display of functional, full-length human and viral membrane proteins. Bioorg Med Chem Lett. 2008 Nov 15;18(22):5937-40. doi: 10.1016/j.bmcl.2008.07.051. Epub 2008 Jul 17. PMID 18667306
- [Background] Levin AM, Weiss GA. Optimizing the affinity and specificity of proteins with molecular display. Mol Biosyst. 2006 Jan;2(1):49-57. doi: 10.1039/b511782h. Epub 2005 Nov 8. PMID 16880922
- [Background] Davis MI, Bennett MJ, Thomas LM, Bjorkman PJ. Crystal structure of prostate-specific membrane antigen, a tumor marker and peptidase. Proc Natl Acad Sci U S A. 2005 Apr 26;102(17):5981-6. doi: 10.1073/pnas.0502101102. Epub 2005 Apr 18. PMID 15837926
- [Background] Hajduczki A, Majumdar S, Fricke M, Brown IA, Weiss GA. Solubilization of a membrane protein by combinatorial supercharging. ACS Chem Biol. 2011 Apr 15;6(4):301-7. doi: 10.1021/cb1001729. Epub 2011 Jan 14. PMID 21192634
- [Background] Lunder, M., Bratkovic, T., Anderluh, G., Strukelj, B., and Kreft, S. (2008) Affinity ranking of phage-displayed peptides: Enzyme-linked immunosorbent assay versus surface plasmon resonance, Acta Chimica Slovenica 55, 233-235.
- [Background] Murase K, Morrison KL, Tam PY, Stafford RL, Jurnak F, Weiss GA. EF-Tu binding peptides identified, dissected, and affinity optimized by phage display. Chem Biol. 2003 Feb;10(2):161-8. doi: 10.1016/s1074-5521(03)00025-5. PMID 12618188
- [Background] Weiss GA, Watanabe CK, Zhong A, Goddard A, Sidhu SS. Rapid mapping of protein functional epitopes by combinatorial alanine scanning. Proc Natl Acad Sci U S A. 2000 Aug 1;97(16):8950-4. doi: 10.1073/pnas.160252097. PMID 10908667
- [Background] Avrantinis SK, Stafford RL, Tian X, Weiss GA. Dissecting the streptavidin-biotin interaction by phage-displayed shotgun scanning. Chembiochem. 2002 Dec 2;3(12):1229-34. doi: 10.1002/1439-7633(20021202)3:123.0.CO;2-X. PMID 12465031
- [Background] Mohan K, Weiss GA. Dual genetically encoded phage-displayed ligands. Anal Biochem. 2014 May 15;453:1-3. doi: 10.1016/j.ab.2014.02.025. Epub 2014 Mar 4. PMID 24607794
- [Background] Levin AM, Murase K, Jackson PJ, Flinspach ML, Poulos TL, Weiss GA. Double barrel shotgun scanning of the caveolin-1 scaffolding domain. ACS Chem Biol. 2007 Jul 20;2(7):493-500. doi: 10.1021/cb700055t. Epub 2007 Jun 29. PMID 17602618
- [Background] Levin AM, Coroneus JG, Cocco MJ, Weiss GA. Exploring the interaction between the protein kinase A catalytic subunit and caveolin-1 scaffolding domain with shotgun scanning, oligomer complementation, NMR, and docking. Protein Sci. 2006 Mar;15(3):478-86. doi: 10.1110/ps.051911706. Epub 2006 Feb 1. PMID 16452625
- [Background] Nutiu R, Li Y. In vitro selection of structure-switching signaling aptamers. Angew Chem Int Ed Engl. 2005 Feb 4;44(7):1061-1065. doi: 10.1002/anie.200461848. No abstract available. PMID 15643624
- [Background] Oh SS, Plakos K, Lou X, Xiao Y, Soh HT. In vitro selection of structure-switching, self-reporting aptamers. Proc Natl Acad Sci U S A. 2010 Aug 10;107(32):14053-8. doi: 10.1073/pnas.1009172107. Epub 2010 Jul 26. PMID 20660786
- [Background] Tuerk C, Gold L. Systematic evolution of ligands by exponential enrichment: RNA ligands to bacteriophage T4 DNA polymerase. Science. 1990 Aug 3;249(4968):505-10. doi: 10.1126/science.2200121.
- [Background] Ellington AD, Szostak JW. In vitro selection of RNA molecules that bind specific ligands. Nature. 1990 Aug 30;346(6287):818-22. doi: 10.1038/346818a0. PMID 1697402
- [Background] Liu J, Cao Z, Lu Y. Functional nucleic acid sensors. Chem Rev. 2009 May;109(5):1948-98. doi: 10.1021/cr030183i. No abstract available. PMID 19301873
- [Background] Zhao W, Ali MM, Aguirre SD, Brook MA, Li Y. Paper-based bioassays using gold nanoparticle colorimetric probes. Anal Chem. 2008 Nov 15;80(22):8431-7. doi: 10.1021/ac801008q. Epub 2008 Oct 11. PMID 18847216
- [Background] Wood JB, Szyndler MW, Halpern AR, Cho K, Corn RM. Fabrication of DNA microarrays on polydopamine-modified gold thin films for SPR imaging measurements. Langmuir. 2013 Aug 27;29(34):10868-73. doi: 10.1021/la402425n. Epub 2013 Aug 15. PMID 23902428
- [Background] Toma M, Loget G, Corn RM. Flexible Teflon nanocone array surfaces with tunable superhydrophobicity for self-cleaning and aqueous droplet patterning. ACS Appl Mater Interfaces. 2014 Jul 23;6(14):11110-7. doi: 10.1021/am500735v. Epub 2014 Apr 1. PMID 24654844